CLINICAL TRIAL: NCT04947267
Title: To Compare the Pulpal Oxygen Saturation Level After Administering Mepivacaine With and Without Vasoconstrictor: A Randomized Clinical Trial
Brief Title: To Compare the Pulpal Oxygen Saturation Level After Administering Mepivacaine With and Without Vasoconstrictor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afshan Amjad Ali (Other)
Responsible Party: Sponsor-Investigator, Afshan Amjad Ali, Principal Investigator, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: AAAli
Record Dates: First submitted 2021-06-18; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: LOCAL ANESTHESIA
Keywords: pulpal oxygen saturation
MeSH Terms: interventions — Mepivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2 % MEPIVACAINE WITH 1:100,000 EPINEPHRINE AND 3% MEPIVACAINE BOTH WERE MASKED BY DENTAL ASSISTANT WITH PINK AND BLUE COLOR RESPECTIVELY.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3% mepivacaine (Experimental): 3% mepivacaine was administered via inferior alveolar nerve block.
  Interventions: Drug: 3% Mepivacaine Hydrochloride
- 2% mepivacaine with 1:100,000 epinephrine (Active Comparator): 2% mepivacaine with 1:100,000 epinephrine was administered via inferior alveolar nerve block.
  Interventions: Drug: 2% Mepivacaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 3% Mepivacaine Hydrochloride — 1.8 ml of 3% mepivacaine (3% Scandonest, Septodont) was administered to Group B patients. Inferior alveolar nerve block was administered to both the groups. Rubber dam was then placed in the desired quadrant. Selected carious mandibular was restored and seven pulpal oxygen saturation spot readings were taken for an hour.
  Other Names: 3% scandonest plain
  Arms: 3% mepivacaine
Drug: 2% Mepivacaine with 1:100,000 epinephrine — 1.8 ml of 2% mepivacaine with 1:100,000 epinephrine (2% Scandonest Special, Septodont) was administered to Group A patients. Inferior alveolar nerve block was administered to both the groups. Rubber dam was then placed in the desired quadrant. Selected carious mandibular was restored and seven pulpal oxygen saturation spot readings were taken for an hour.
  Other Names: 2% scandonest special
  Arms: 2% mepivacaine with 1:100,000 epinephrine

SUMMARY:
As vasoconstrictors adversely affect pulpal hemodynamics, this study compared the pulpal oxygen saturation levels after employing inferior alveolar nerve block with 2% mepivacaine with 1:100,000 epinephrine (2% Scandonest Special) and 3% mepivacaine (3% Scandonest Plain).Two groups were made with 30 patients in each group. 2% mepivacaine with 1:100,000 epinephrine (2% Scandonest Special) was administered to the patients in Group A whereas 3% mepivacaine (3% Scandonest Plain) was administered to the patients in Group B. Rubber dam application, cavity preparation and composite filling was then done on the selected carious mandibular premolar. Pulpal oxygen saturation levels were recorded after administration of local anesthesia with Nellcor-550 pulse oximeter and Nellcor D-YS Multisite reusable sensor.

DETAILED DESCRIPTION:
BACKGROUND ' Local anesthesia is the foremost requirement of an efficient operative dental procedure to be executed in a pain free and calm environment. Local anesthesia is available in two forms: with vasoconstrictor and without vasoconstrictor. As vasoconstrictors adversely affect pulpal hemodynamics, this study aims to compare the pulpal oxygen saturation levels after employing inferior alveolar nerve block with 2% mepivacaine with 1:100,000 epinephrine (2% Scandonest Special) and 3% mepivacaine (3% Scandonest Plain).

NULL HYPOTHESIS There is no difference between the pulpal oxygen saturation levels after administering 2% mepivacaine with 1:100,000 epinephrine and 3% mepivacaine.

ALTERNATE HYPOTHESIS There is a difference between the pulpal oxygen saturation levels after administering 2% mepivacaine with 1:100,000 epinephrine and 3% mepivacaine.

METHOD Two groups were made with 30 patients in each group. 2% mepivacaine with 1:100,000 epinephrine (2% Scandonest Special) was administered to the patients in Group A whereas 3% mepivacaine (3% Scandonest Plain) was administered to the patients in Group B. Rubber dam application, cavity preparation and composite filling was then done on the selected carious mandibular premolar. Pulpal oxygen saturation levels were recorded after administration of local anesthesia with the Nellcor- PM 10N pulse oximeter and Nellcor D-YS Multisite reusable sensor.

STATISTICAL ANALYSIS The statistical package for social sciences version 21.0 is used for statistical analysis. Mean and standard deviation of the pulpal oxygen saturation levels for filled and unfilled teeth under the effect of 2% mepivacaine with 1:100,000 epinephrine and 3% mepivacaine were recorded. Mixed Way ANOVA will be applied to discern if there is any difference in the pulpal oxygen saturation levels within and between the two groups. Post Hoc Tuckey was applied to identify whether the paired difference is present within groups or between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Medical status: healthy individuals with no current and past medical findings.
* Medications: no current medications.
* Both mature vital ipsilateral mandibular premolars:

  * Healthy premolar (ICDAS code 0)
  * Carious premolar (ICDAS code 4-6).
* Periapical status

  * Healthy premolar - Periapical Index. (Code 1).
  * Carious premolar - Periapical Index. (Code 1).
* Periodontal status

  * Healthy premolar - Classification of periodontal diseases and conditions (Code 0).
  * Carious premolar - Classification of periodontal diseases and conditions (Code 0).

Exclusion Criteria:

* Patients with oral and maxillofacial syndromes and anomalies.
* Pregnant and nursing mothers.
* Class V carious lesions (sensor of pulse oximeter was placed on intact buccal, lingual and cervical surfaces).
* Teeth with extracoronal restorations.
* Teeth with developmental defects and other anomalies.
* Dental trauma.
* Teeth with symptoms of irreversible pulpitis.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
PULPAL OXYGEN SATURATION | 60 minutes
  Pulpal oxygen saturation levels were recorded for 60 min after administration of local anesthesia using Nellcor-PM10N pulse oximeter and Nellcor D-YS Multisite reusable sensor.

CONTACTS AND LOCATIONS:
Overall Officials: AFSHAN AMJAD ALI, MSc, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No